CLINICAL TRIAL: NCT06667219
Title: Influencing Factors and Interventions of Physical Exercise Behaviour of 6-Year-Old Children in Guangdong, China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Zhang Haiyan, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: USM/JEPeM/KK/23030260
Record Dates: First submitted 2024-10-24; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-04

CONDITIONS: Physical Exercise Behaviour; Fundamental Motor Skills; 6-Year-Old Children
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Children will be invited to participate in the after-school physical activity experiment.This experiment will include more than 108 participants randomly assigned to the experimental group (n=54) and the control group (n=54) (randomly selected two kindergartens, one as experimental group and one as control group). All studies will be conducted in Zengcheng Kindergarten, Guangdong, China. Children will participate in this study and participats (parents/guardians) will receive a prescription for childhood exercise.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group, a children's physical fitness training program (Experimental): Length:12 weeks, 40 minutes one time, twice a week.
  Intervention content:
  The intervention will be conducted using a relevant physical fitness training program.
  Interventions: Behavioral: A relevant physical fitness training program intervention
- control group, Physical exercise using kindergarten standards (Experimental): Duration: 12 weeks. Content: Physical exercise using kindergarten standards.
  Interventions: Behavioral: control group,Physical exercise using kindergarten standards

INTERVENTIONS:
Behavioral: A relevant physical fitness training program intervention — 54children who participated in after-school sports activities in Guangzhou Kindergarten (Guangzhou, China) were randomly selected as the experimental group.
  Intervention group Length:12 weeks, 40 minutes, twice a week.
  Intervention content:
  The intervention will be conducted using a relevant physical fitness training program , as follows: Week 1 / 4 first: Run quickly;Durian ball;Throw;Fast jogging (200 m) Week 1 / 4 second: Dodge run,Raise your legs high and go over the small hurdles; Durian ball (standing on one foot);standing long jump Week 2 / 5 first: Bow step transformation jump;Throw;Turn back 10 meters Week 2 / 5 second: Hop ;Stand on one foot with your eyes open Week 3 / 6 first:Skip over the small hurdles;Durian ball (standing on one foot);Throw; Fast jogging (200 m) Week 3 / 6 second:Jump on your feet and dodge running;Durian ball (squat);Jump support Weeks 7-12,Repeat the above content. FMS index was tested before the experiment, and once after the intervention.
  Arms: Intervention group, a children's physical fitness training program
Behavioral: control group,Physical exercise using kindergarten standards — 54 children who did not participate in after-school sports activities were selected as the control group.
  control group Duration: 12 weeks. Content: Physical exercise using kindergarten standards. FMS index was tested the same to intervention group before the test and FMS index was measured once again after 12 weeks.
  Arms: control group, Physical exercise using kindergarten standards

SUMMARY:
The goal of this clinical trial is to examine the relationship between children's physical exercise behavior and children's Fundamental Motor Skills (FMS) before and after changing the influencing factors of 6-year-old children's physical exercise behavior in Guangdong Province, China. The main question it aims to answer is:

Is there any change of the relationship (time, group, and interaction) between 6-year-old children's physical exercise behaviour and children's Fundamental Motor Skills (FMS) before and after the physical activity intervention of the influencing factors in Guangdong Province, China?

Participants will:

Intervention group, Length: 12 weeks, 40 minutes, twice a week. The intervention will be conducted using a relevant physical fitness training program.

Control group, Length: 12 weeks. Content: Physical exercise using kindergarten standards.

Researchers will compare the data before and after the intervention to know whether the Fundamental Motor Skills (FMS) of 6-year-old children have changed.

ELIGIBILITY:
Inclusion Criteria:

* Preschool children aged 6 years old in Guangdong, China;
* Children who are of Chinese nationality;
* Male and female;
* Parents/guardians signed an informed consent form;

Exclusion Criteria:

* Have a mental illness with cognitive impairment problems;
* Children with speech or ear function impairment;
* Recent or imminent surgery (within 3 months), or medical co-morbidities;
* Parents/guardians did not sign the informed consent.

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2024-08-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Changes in test values of 13 indicators of Fundmental Motor Skills in 6-year-old children at 12 weeks | 5 months
  The FMS is measured with the tool TGMD-3. TGMD-3 is scored based on the completion quality of children.
  The unit of measurement is "scores". The 13-item test consists of two subscales: six locomotor skills (LM) (i.e., run, gallop, hop, slide, jump, and skip) and seven ball skills (BS), formerly known as object control skills (i.e., forehand strike, two-hand strike, overhand throw, underhand throw, dribble, catch, and kick). According to the TGMD-3, each skill has a set of performance criteria that is evaluated. In this case, raw scores for locomotor skills could range from 0 to 46. Similarly, ball skills could range from 0 to 54. The total score of all movements was 100 scores.
  The higher score represents a higher level of motor skill development, and the low score indicates a lack of some critical movement development.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Huali College, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No